CLINICAL TRIAL: NCT01431222
Title: Interventional Strategy to Abrogate Mitral Regurgitation Using the MitraClip System in High-Risk Patients Considered Unsuitable for Surgery (ISAR-CLIP)
Brief Title: Abrogation of Mitral Regurgitation Using the MitraClip System in High-Risk Patients Unsuitable for Surgery
Acronym: ISAR-CLIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Joerg Hausleiter, Klinik für Herz- und Kreislauferkrankungen, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IsarClip
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Mitral Regurgitation
Keywords: severe mitral regurgitation; interventional mitral valve reconstruction; inoperable; EuroSCORE; STS Risk Score; MitraClip; fluoroscopy; echocardiography; percutaneous treatment of mitral regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- percutaneous treatment (Active Comparator)
  Interventions: Device: percutaneous treatment by implanting a Mitra Clip device
- optimal medical treatment (No Intervention)
  Interventions: Device: percutaneous treatment by implanting a Mitra Clip device

INTERVENTIONS:
Device: percutaneous treatment by implanting a Mitra Clip device — With a minimal-invasive, percutaneous catheter-based technique and trans-septal approach under transesophageal echocardiographic and fluoroscopic guidance, the MitraClip device grasps and approximates the mitral leaflets thus creating a double-orifice mitral valve with a permanent leaflet coaptation and a reduction or even abrogation of mitral regurgitation.
  Other Names: Mitra Clip system

SUMMARY:
The primary objective in this randomized trial is to evaluate the safety and efficacy of a MitraClip treatment in symptomatic patients with severe mitral regurgitation in comparison to the previous default medical treatment - in a study population who is not amenable for the conventional surgical approach as current gold standard.

DETAILED DESCRIPTION:
The presence of a significant mitral regurgitation (MR) seriously effects the patient's quality of life and is associated with an increased mortality rate. The operative treatment of MR - either mitral valve repair or replacement - is the current gold standard. However mere half of the patients with a severe and symptomatic MR actually undergo an operative treatment (EURO-HEART-SURVEY) due to restricted left ventricular ejection fraction, elderly patients with co-morbidities and high perioperative morbidity and mortality. In contrast, patients with severe and symptomatic MR not suitable for operation are treated with palliative medical therapy (heart insufficiency therapy). With the development of the MitraClip device - a minimal-invasive, percutaneous catheter-based technique - high-risk patients not suitable for surgery may receive a promising alternative treatment by approximating the mitral leaflets, thus creating a permanent leaflet coaptation and reducing or even abrogating the MR. The current data support the assumption of a safe and effective MR reduction with the MitraClip-System in inoperable high-risk patients with severe MR. But the feasibility still has to be proven in this special patient population.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* signed written consent
* symptomatic patients (NYHA-stadium ≥ III) for at least 3 months with an exploited medical heart insufficiency therapy
* increased perioperative risk with a logistic EuroScore ≥ 15 or STS-Score ≥ 15
* MR grade ≥ 2, amenable for MitraClip intervention assessed by an experienced interventional cardiologist
* Affirmation of in-operability by a "Heart-Team" consisting of either 1 cardiac surgeon and 1 cardiologist or 3 cardiologists

Exclusion Criteria:

* one essential cardiovascular event in the past 6 weeks; i. e. myocardial infarction, stroke, shock, cardiac decompensation, or the necessity of catecholamine therapy for haemodynamic stabilisation
* implantation of a biventricular pacemaker-device for cardiac resynchronisation therapy in the past 3 months
* solid tumor with a live expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of Dyspnoea of at least one class (NYHA-Classification) | after 6 months

SECONDARY OUTCOMES:
composite endpoint and clinical outcome measured by NYHA-classification | 1 year and 2 years after intervention
  * composite endpoint (death of any cause, myocardial infarction, stroke, sepsis, TIMI major bleeding, clip embolisation, partial clip detachement, acute renal failure)
  * unscheduled hospitalization due to increased heart insuffiecency
  * changes in quality of life
  * echocardiographic parameters
  * loboratory parameters
  * resiliance measured by spiroergometry

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, MD, Study Chair — Deutsches Herzzentrum Muenchen; Steffen Massberg, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Juergen Pache, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Hasema Lesevic, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Bavaria, Germany